CLINICAL TRIAL: NCT06787820
Title: Evaluation of the Cognitive and Socioemotional Impact of a Musical Intervention in Older Adults
Brief Title: Impact of a Musical Intervention in Older Adults (ARA Project - Armonía Recreativa Para El Adulto Mayor)
Acronym: ARA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Diego Portales (Other)
Responsible Party: Principal Investigator, Leonie Kausel, Principal Investigator, University Diego Portales
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDP 01-2024; Fondo Académicas Res 150/2023 (Other Grant/Funding Number: Universidad Diego Portales, Chile)
Record Dates: First submitted 2025-01-03; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-06

CONDITIONS: Older People
Keywords: Music; Elderly persons; Institutionalized
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Control: Participants will attend concerts held within the care facility
  Experimental: Group musical intervention once a week in 60-minute sessions for three months, a sufficient duration to observe changes (Mathew et al., 2017). Sessions will be designed by the principal investigator and a music teacher, and conducted by the experienced music teacher. Activities will include experiencing sound qualities (pitch, duration, intensity, and timbre) through movement, with a focus on collective participation and learning. Musical preferences of participants will be considered in the session design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music intervention (Experimental): Group musical intervention once a week in 60-minute sessions for three months, a sufficient duration to observe changes (Mathew et al., 2017). Sessions will be designed by the principal investigator and a music teacher, and conducted by the experienced music teacher. Activities will include experiencing sound qualities (pitch, duration, intensity, and timbre) through movement, with a focus on collective participation and learning. Musical preferences of participants will be considered in the session design.
  Interventions: Behavioral: Music intervention
- Listen to music (No Intervention): Participants will attend three concerts, one per month, held within the care facility

INTERVENTIONS:
Behavioral: Music intervention — The musical intervention conducted at the senior home focused on the development of rhythmic and vocal skills, as well as the creation of educational experiences that promoted the acquisition of these competencies. To achieve this, both conventional percussion instruments, such as claves, tambourines, woodblocks, and triangles, and unconventional elements, such as buckets played with drumsticks, sheets of paper, spoons, ribbons, elastic bands, and a parachute, were used to mark the rhythm during the singing sessions. The selected songs were chosen based on the musical styles mentioned by the participants during the pre-intervention interview. Furthermore, participants were given the opportunity to showcase their progress at the end of the activity, with the aim of sharing these achievements with family and friends at the home.
  Other Names: Music therapy
  Arms: Music intervention

SUMMARY:
Currently, the world is facing the challenge of population aging. At this stage of life, various deteriorations, such as cognitive decline, begin to appear, significantly impairing the quality of life. Therefore, it is imperative to seek interventions that can positively impact the life trajectory of older adults. While the cognitive benefits of musical interventions for children and young people are well-documented, there is a lack of evidence regarding their effects on the cognitive and socioemotional well-being of institutionalized older adults.

To address this, the investigators will conduct a non-randomized clinical trial at Fundación Las Rosas, which operates various homes for the elderly. The trial will involve two groups: a control group and an experimental group. The control group will attend concerts held within the care facility, while the experimental group will participate in a music workshop once a week for three months.

To evaluate the outcomes, cognitive and socioemotional assessments will be conducted at three points: prior to the musical intervention (baseline), at the end of the intervention period, and one month after the interventions conclude (follow-up). The results will provide valuable insights to support the development and implementation of cost-effective non-pharmacological interventions, specifically musical interventions, to promote well-being in older adults by demonstrating their applicability and effectiveness within the national context. By assessing the intervention's impact on both cognitive and socioemotional dimensions, this study will also contribute to a deeper understanding of how these skills can be developed and promoted among older adults.

DETAILED DESCRIPTION:
The world is facing a gradual aging of the population. It is estimated that in the coming years, people over 60 years old will outnumber children under 10 years old, and by 2050, the population over 60 will surpass adolescents and young adults worldwide. Additionally, the population of those over 80 years old is expected to triple by 2050. Chile is also following this global trend. This reality underscores the need to understand how to ensure well-being during this life stage is not diminished by natural aging processes and their context, such as cognitive decline or the weakening of socioemotional well-being.

Music has been a form of expression accompanying humans since ancient times. It is a powerful generator of emotions , evocative of memories, and a creator of social cohesion. Importantly, it has shown positive effects on both cognitive and socioemotional aspects when musical interventions are implemented in older adults, in both clinical cases and typical aging. Active musical interventions include activities such as singing, playing an instrument, and/or moving to the rhythm of the music. The success of these interventions is proposed to be due to their requirements for multisensory integration, cognitive demands, promotion of social interaction and bond formation, perception as enjoyable and entertaining, and inherent motivational qualities that evoke positive emotions. These types of interventions could be highly relevant in the national context, for example, for the "Active Aging" program of the National Service for the Elderly (SENAMA) of the Ministry of Social Development and Family, which seeks to have self-sufficient older adults participate in activities that promote active aging, as well as for the National Comprehensive Health Plan for Older Adults, which proposes a series of actions framed, among other things, in the prevention of health problems. Therefore, it is urgent to evaluate the effectiveness of these interventions in our sociocultural context, particularly in nursing homes where residents often lack an extended network to care for them, making these interventions particularly important for those in vulnerable situations, and where such interventions have shown positive impacts.

This study proposes to evaluate the impact on both cognitive and socioemotional dimensions of a musical intervention in institutionalized older adults. Importantly, a study is proposed in which the participating institutions will be randomized to either the intervention group, where older adults will receive the musical intervention, or the control group, where they will not receive the intervention, following current recommendations for evaluating the impact of musical interventions in prevention and rehabilitation contexts. Evaluations of cognitive functions and socioemotional well-being will be conducted at three time points for both groups: baseline pre-intervention, post-intervention immediately after the intervention concludes, and follow-up one month after the intervention concludes. This design will elucidate the effect of the musical intervention on older adults and the persistence of these changes. The results of this study will be a starting point to promote research on musical interventions focused on the well-being of the older population in Chile. Additionally, they will allow applications for funding to continue investigating the most effective forms of intervention for this age group and understanding the mechanisms by which these interventions act, for example, using neurobiological activity measurement techniques from neuroscience.

General Aim

To evaluate the impact on cognitive and socioemotional dimensions of a musical intervention in older adults residing in a nursing home.

Specific Aim

1. To determine changes in cognitive functions and socioemotional well-being pre- and post-musical intervention in both the intervention and control groups.
2. To assess the persistence of cognitive and socioemotional changes post-intervention in both groups.
3. To analyze similarities and differences in cognitive functions and socioemotional well-being across all evaluation stages (pre, post, follow-up) between the intervention and control groups.

Methods

A non-randomized clinical study, quasi-experimental in nature, will be conducted, recording changes at three time points: a) pre-intervention, b) post-intervention, and c) follow-up.

Senior citizen Residences The study will take place at Fundación Las Rosas in Santiago, Chile. Each participant will be individually invited and informed about the study, with all consent points reviewed in a conducive environment for uninterrupted conversation.

Interventions

* Control:** Participants will attend concerts held within the care facility
* Experimental:** Group musical intervention once a week in 60-minute sessions for three months, a sufficient duration to observe changes (Mathew et al., 2017). Sessions will be designed by the principal investigator and a music teacher, and conducted by the experienced music teacher. Activities will include experiencing sound qualities (pitch, duration, intensity, and timbre) through movement, with a focus on collective participation and learning. Musical preferences of participants will be considered in the session design.

Evaluations and outcomes

Evaluations of cognitive and socioemotional functioning will be assessed three times: 1) at baseline, prior to the musical intervention; 2) post-intervention, immediately after the intervention concludes; and 3) follow up, one month after the intervention concludes.

During the second evaluation (post-intervention), a Satisfaction Survey will also be administered to the intervention group to gauge acceptance and feedback for refining the intervention.

This study aims to enhance understanding of the effects of musical interventions on older adults and provide valuable data to develop more effective programs, ultimately improving the quality of life for the elderly population in Chile.

ELIGIBILITY:
Inclusion Criteria:

* Older adults residing in a protected residence.
* Consent to participate in the study.

Exclusion Criteria:

* Physical or cognitive impairments that prevent participation in musical intervention activities.
* Mild cognitive impairment determined by the GDS-3 scale, reported by the residence therapists.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive performance - Montreal Cognitive Assessment (MoCA) | These assessments will be administered three times: 1) at baseline, prior to the musical intervention; 2) immediately after the intervention concludes; and 3) follow up, one month after the intervention concludes.
  Montreal Cognitive Assessment (MoCA). This is a screening test that provides a comprehensive evaluation of global cognition and various cognitive functions. Values range from 0 - 30, with a higher score meaning a better outcome.
Cognitive performance - Phototest | These assessments will be administered three times: 1) at baseline, prior to the musical intervention; 2) immediately after the intervention concludes; and 3) follow up, one month after the intervention concludes.
  Phototest. A brief cognitive screening test applicable to illiterate people that through the recognition and naming of images of everyday objects offers insights into facilitated memory, denomination and verbal fluency. It can be used for the detection of cognitive impairment and dementia. Values range from 0 on, because the maximum value depends on how many objects the person recognizes or names. Higher scores mean a better outcome, and a score of 28 or less is an indicator of cognitive decline.
Cognitive performance - Test of Executive Functions Free from Schooling Bias (TELE) | These assessments will be administered three times: 1) at baseline, prior to the musical intervention; 2) immediately after the intervention concludes; and 3) follow up, one month after the intervention concludes.
  Test of Executive Functions Free from Schooling Bias (TELE, Test de funciones Ejecutivas Libre de sesgo por Escolaridad).
  The TELE consists of an executive function evaluation task that screens inhibitory control, sustained attention, verbal working memory and processing speed. Values range from 0 - 12, where higher scores mean a better outcome.
Socioemotional performance - UCLA Loneliness Scale | These assessments will be administered three times: 1) at baseline, prior to the musical intervention; 2) immediately after the intervention concludes; and 3) follow up, one month after the intervention concludes.
  University of California Los Angeles Loneliness Scale (UCLA Loneliness Scale). A scale to detect the feeling of loneliness through 10 questions that score between 1 and 4 points, allowing a minimum score of 10 and a maximum of 40. Higher scores mean a better outcome.
Socioemotional performance - Geriatric Depression Scale (GDS) | These assessments will be administered three times: 1) at baseline, prior to the musical intervention; 2) immediately after the intervention concludes; and 3) follow up, one month after the intervention concludes.
  Geriatric Depression Scale (GDS). This is a self-report instrument composed of 30 items that measure the presence of depressive symptomatology through direct questions, 20 of which measure the presence of symptoms ("Do you feel that your life is empty?"), while 10 are considered inverse items ("Are you basically satisfied with your life?"). It is a dichotomous scale in which the respondent answers yes or no. The scores range from 0 - 30, where high scores indicate a worse outcome, suggesting high risks of depression.

SECONDARY OUTCOMES:
Functionality performance - Activities of Daily Living Questionnaire (ADLQ) | These assessments will be administered three times: 1) at baseline, prior to the musical intervention; 2) immediately after the intervention concludes; and 3) follow up, one month after the intervention concludes.
  Activities of Daily Living Questionnaire (ADLQ). This questionnaire asks about functionality in every day life activities, using a 4-point scale to measure functional capacity. The score ranges from 0 - 100, where higher scores indicate a worse outcome, suggesting higher risks of significant functional impairment in daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Las Rosas, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Carnero-Pardo C, Montoro-Rios MT. [The photo test]. Rev Neurol. 2004 Nov 1-15;39(9):801-6. Spanish. PMID 15543492
- [Background] Caldichoury N, Soto-Anari M, Camargo L, Porto MF, Herrera-Pino J, Shelach S, Rivera-Fernandez C, Ramos-Henderson M, Gargiulo PA, Lopez N. Clinical utility of Phototest via teleneuropsychology in Chilean rural older adults. Dement Neuropsychol. 2022 Jul-Sep;16(3):316-323. doi: 10.1590/1980-5764-DN-2021-0082. Epub 2022 Jun 24. PMID 36619838
- [Background] Law LN, Zentner M. Assessing musical abilities objectively: construction and validation of the profile of music perception skills. PLoS One. 2012;7(12):e52508. doi: 10.1371/journal.pone.0052508. Epub 2012 Dec 28. PMID 23285071
- [Background] Velarde-Mayol C, Fragua-Gil S, Garcia-de-Cecilia JM. [Validation of the UCLA loneliness scale in an elderly population that live alone]. Semergen. 2016 Apr;42(3):177-83. doi: 10.1016/j.semerg.2015.05.017. Epub 2015 Jul 14. Spanish. PMID 26187595
- [Background] Abraha I, Rimland JM, Trotta FM, Dell'Aquila G, Cruz-Jentoft A, Petrovic M, Gudmundsson A, Soiza R, O'Mahony D, Guaita A, Cherubini A. Systematic review of systematic reviews of non-pharmacological interventions to treat behavioural disturbances in older patients with dementia. The SENATOR-OnTop series. BMJ Open. 2017 Mar 16;7(3):e012759. doi: 10.1136/bmjopen-2016-012759. PMID 28302633
- [Background] Boer D, Abubakar A. Music listening in families and peer groups: benefits for young people's social cohesion and emotional well-being across four cultures. Front Psychol. 2014 May 8;5:392. doi: 10.3389/fpsyg.2014.00392. eCollection 2014. PMID 24847296
- [Background] Edwards E, St Hillaire-Clarke C, Frankowski DW, Finkelstein R, Cheever T, Chen WG, Onken L, Poremba A, Riddle R, Schloesser D, Burgdorf CE, Wells N, Fleming R, Collins FS. NIH Music-Based Intervention Toolkit: Music-Based Interventions for Brain Disorders of Aging. Neurology. 2023 May 2;100(18):868-878. doi: 10.1212/WNL.0000000000206797. Epub 2023 Jan 13. PMID 36639235
- [Background] Grau-Sanchez J, Jamey K, Paraskevopoulos E, Dalla Bella S, Gold C, Schlaug G, Belleville S, Rodriguez-Fornells A, Hackney ME, Sarkamo T. Putting music to trial: Consensus on key methodological challenges investigating music-based rehabilitation. Ann N Y Acad Sci. 2022 Dec;1518(1):12-24. doi: 10.1111/nyas.14892. Epub 2022 Sep 30. PMID 36177875
- [Background] Juslin PN, Vastfjall D. Emotional responses to music: the need to consider underlying mechanisms. Behav Brain Sci. 2008 Oct;31(5):559-75; discussion 575-621. doi: 10.1017/S0140525X08005293. PMID 18826699
- [Background] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Background] Sarkamo T. Cognitive, emotional, and neural benefits of musical leisure activities in aging and neurological rehabilitation: A critical review. Ann Phys Rehabil Med. 2018 Nov;61(6):414-418. doi: 10.1016/j.rehab.2017.03.006. Epub 2017 Apr 29. PMID 28461128
- [Background] Sihvonen AJ, Sarkamo T, Leo V, Tervaniemi M, Altenmuller E, Soinila S. Music-based interventions in neurological rehabilitation. Lancet Neurol. 2017 Aug;16(8):648-660. doi: 10.1016/S1474-4422(17)30168-0. Epub 2017 Jun 26. PMID 28663005
- [Background] Stietz J, Pollerhoff L, Kurtz M, Li SC, Reiter AMF, Kanske P. The ageing of the social mind: replicating the preservation of socio-affective and the decline of socio-cognitive processes in old age. R Soc Open Sci. 2021 Aug 25;8(8):210641. doi: 10.1098/rsos.210641. eCollection 2021 Aug. PMID 34457343
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Heinze HG, Bohn U. [Iodine-131 therapy of autonomous adenoma of the thyroid. 7-year results]. Dtsch Med Wochenschr. 1987 Jul 3;112(27):1073-9. doi: 10.1055/s-2008-1068196. German. PMID 3595467
- [Background] Zhang Y, Cai J, An L, Hui F, Ren T, Ma H, Zhao Q. Does music therapy enhance behavioral and cognitive function in elderly dementia patients? A systematic review and meta-analysis. Ageing Res Rev. 2017 May;35:1-11. doi: 10.1016/j.arr.2016.12.003. Epub 2016 Dec 23. PMID 28025173